CLINICAL TRIAL: NCT06671509
Title: A Phase 1 Open-Label Single-Dose Study to Assess the Pharmacokinetics and Safety of YZJ-1139 in Subjects With Mild, Moderate and Normal Hepatic Impairment
Brief Title: Pharmacokinetics and Safety Study of YZJ-1139 in Subjects With Mild, Moderate and Normal Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Haiyan Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZJ-1139-1-11
Record Dates: First submitted 2024-11-01; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Insomnia; Hepatic Impairment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Single dose
Masking Description: Non-randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Mild Hepatic Impairment (Experimental)
  Interventions: Drug: YZJ-1139
- Group B: Moderate Hepatic Impairment (Experimental)
  Interventions: Drug: YZJ-1139
- Group C: Normal Hepatic Impairment (Experimental)
  Interventions: Drug: YZJ-1139

INTERVENTIONS:
Drug: YZJ-1139 — Single oral dose, 20 mg tablet

SUMMARY:
Primary Objectives:

To evaluate the effect of the subjects with mild (Child Pugh A), moderate (Child Pugh B) and normal hepatic impairment on the pharmacokinetics of YZJ-1139

Secondary Objectives:

To evaluate the safety of a single oral dose of YZJ-1139 in subjects with mild, moderate and normal hepatic impairment

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form before the start of activities related to this trial, and be able to understand the procedures and methods of this trial, willing to strictly follow the clinical trial protocol to complete this trial;
2. The subjects (including partners) are willing to self screen and have no family planning within 3 months after the administration of the investigational drug, and voluntarily take contraceptive measures (see Appendix 1 for specific contraceptive measures);
3. On the day of signing the informed consent form, the age range is 18 to 70 years old (including both ends), both men and women are eligible;
4. The weight of male subjects shall not be less than 50 kg, and the weight of female subjects shall not be less than 45 kg; Body mass index (BMI) 18-32 kg/m2 (including both ends);
5. Creatinine clearance rate (calculated using Cockcroft Gault formula, see Appendix 2) ≥ 60 mL/min;

   Subjects with liver dysfunction also need to meet all the following conditions:
6. Chronic liver injury caused by primary liver diseases (such as hepatitis B, hepatitis C, autoimmune hepatitis, alcoholic liver disease, etc.) or clinically diagnosed as cirrhosis (see Appendix 3 for diagnostic criteria for cirrhosis), and liver dysfunction patients with Child Pugh grading of A or B (see Appendix 4 for Child Pugh grading).
7. Individuals who have a stable medication regimen for the treatment of liver dysfunction, complications, and other accompanying diseases for at least 14 days prior to taking the investigational drug, and whose medication does not need to be adjusted (including medication type, dosage, or frequency); Or those who have not taken medication;

   Subjects with normal liver function also need to meet all the following conditions:
8. The demographic mean of subjects in the normal liver function group (Group C) during screening must meet the following matching criteria:

   1. Match the weight with the liver function impairment group (Group A+Group B), with a mean of ± 10 kg;
   2. Age matched with the liver function impairment group (Group A+Group B), with a mean of ± 10 years;
   3. Match with the liver function impairment group (Group A+Group B) by gender, with a mean of ± 1 case;

Exclusion Criteria:

1. Allergic constitution, such as those with a known history of allergies to two or more substances, or those with allergic diseases, or those with a history of allergies to experimental drugs or similar drugs or excipients;
2. Screening period electrocardiogram showed QTc interval (QTcF)>470 msec in males and>480 msec in females (corrected according to Fridericia's standard: QTcF=QT/(RR ^ 0.33), RR=60/heart rate);
3. Screening for individuals who have had severe infections, trauma, gastrointestinal surgery, or other surgical procedures within the first 4 weeks;
4. Individuals with a history of paroxysmal sleep disorder, obstructive sleep apnea, complex sleep behavior (such as dream walking, driving in dreams, etc.), severe unconscious hypoglycemia, stroke, epilepsy, and other psychiatric disorders (including anxiety, depression, etc.), convulsive diseases, and sudden onset of illness;
5. Individuals who have donated blood or lost ≥ 200 mL of blood within the first 3 months of screening, received blood transfusions or used blood products, or planned to donate blood during the trial period or within 1 month after the end of the trial;
6. Individuals who have used CYP3A4 enzyme inducers or inhibitors within one month prior to administration (or five half-lives, whichever is longer) (see Appendix 5);
7. Individuals who have consumed a special diet (including dragon fruit, mango, grapefruit, and/or xanthine diet, chocolate) and/or consumed excessive amounts of tea, coffee, grapefruit/grapefruit juice, and/or caffeinated beverages (an average of 8 or more cups per day, 200mL per cup) within 2 weeks prior to administration;
8. Screening for alcoholics within the first three months, i.e. those who consume more than 14 units of alcohol per week (1 unit ≈ 360 mL of beer, or 45 mL of 40% spirits, or 150 mL of wine) or those who have tested positive for alcohol screening; Screening for individuals who smoke an average of 10 or more cigarettes per day within the first 3 months;
9. Individuals with a history of drug use, drug abuse, or positive drug abuse screening;
10. Pregnant or lactating women, or women who test positive for pregnancy;
11. Patients with difficulty swallowing tablets and special dietary requirements who cannot accept a unified diet;
12. Individuals who cannot tolerate venous puncture or have a history of needle and blood fainting;
13. For other reasons, researchers believe that it is not suitable for inclusion;

    If a subject with liver function impairment meets any of the following exclusion criteria, they need to be excluded:
14. The subject has any of the following conditions: drug-induced liver injury; History of liver transplantation; Cirrhotic patients with liver failure, hepatic encephalopathy, hepatocellular carcinoma (excluding those with Barcelona stage 0 or curative treatment), hepatorenal syndrome, esophageal and gastric variceal bleeding and other complications deemed inappropriate by researchers;
15. Patients with primary biliary cirrhosis and biliary obstruction;
16. The laboratory test results during screening meet any of the following criteria: (a) alanine aminotransferase (ALT) or aspartate aminotransferase (AST)>10 × ULN; (b) Absolute value of neutrophils (NE #)<0.75 × 109/L; (c) Hemoglobin (HGB)<60 g/L; (d) Alpha fetoprotein (AFP)>100 ng/mL;
17. HIV antigen/antibody screening positive individuals; If syphilis antibody is positive, a rapid plasma reactive receptor (RPR) test should be added. If RPR is also positive, it should be excluded;
18. Except for the primary liver disease itself, those who have previously or currently suffered from other serious systemic organ diseases, including but not limited to gastrointestinal, respiratory, renal, neurological, blood, endocrine, tumor, immune, psychiatric or cardiovascular diseases, or clinical laboratory examination abnormalities that are clinically significant and determined by the research doctor to be unsuitable for participation in this trial;
19. Screening for individuals who have used other clinical trial drugs within the first two months or plan to participate in other clinical trials during this study period;

    Subjects with normal liver function who meet any of the following exclusion criteria need to be excluded:
20. Individuals with a history of liver injury;
21. Individuals who have previously or currently suffered from any clinically severe diseases such as circulatory system, endocrine system, nervous system, digestive system, respiratory system, hematology, immunology, psychiatry, and metabolic abnormalities, or any other diseases that can interfere with test results;
22. Abnormal physical examination, vital signs, laboratory tests, 12 lead electrocardiogram, abdominal ultrasound, and other examinations determined by the researcher to have clinical significance;
23. Those who are positive in any index screening of hepatitis B surface antigen, hepatitis C antibody or hepatitis C core antigen, HIV antigen/antibody or syphilis antibody;
24. Those who have used any prescription drugs, over-the-counter drugs, Chinese herbal medicines, or supplements within 14 days before administration;
25. Screening for individuals who have used other clinical trial drugs or plan to participate in other clinical trials during the first three months of this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-04-18 (Actual); Study Completion 2024-08-07 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of YZJ-1139 | From Day 1 to Day 3
  Cmax is defined as the maximum concentration of drug
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUCinf) of YZJ-1139 | From Day 1 to Day 3
  AUCinf is defined as the concentration of drug extrapolated to infinite time
Area Under the Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUClast) of YZJ-1139 | From Day 1 to Day 3
  AUClast is defined as the concentration of drug from time zero to the last observable concentration
Time of Maximum Observed Plasma Concentration (Tmax) of Entrectinib | From Day 1 to Day 3
  Tmax is defined as the time (observed time point) of Cmax.
Apparent Terminal Elimination Half-life (t1/2) of Entrectinib | From Day 1 to Day 3
Apparent Oral Clearance (CL/F) of Entrectinib | From Day 1 to Day 3
  CL/F is defined as the apparent oral clearance following administration of the drug
The Apparent Volume of Distribution (Vz/F) of Entrectinib | From Day 1 to Day 3
  Vz/F is defined as the apparent volume of distribution of the drug

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 to Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China